CLINICAL TRIAL: NCT03429478
Title: Effect of Preoperative Music on "Sterile Inflammation" Induced by Laparoscopic Surgery-A Randomized Study
Brief Title: Effect of Preoperative Music on Sterile Inflammation Induced by Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, PROF. BRIJ B AGARWAL, Vice Chairman Department of General and Laparoscopic Surgery, Sir Ganga Ram Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: EC/10/17/1281
Record Dates: First submitted 2017-11-27; First posted 2018-02-12 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Music Therapy; Cholecystitis/Cholelithiasis; Inflammatory Response; Surgical Injury
Keywords: Music; Laparoscopic Surgery; Sterile Inflammation
MeSH Terms: conditions — Cholecystitis; Cholelithiasis; Intraoperative Complications

STUDY DESIGN:
Intervention Model Description: 50 patients meeting the inclusion criteria will be included in the study after written and informed consent. They will be randomized and divided into 2 groups. Group 1 will be labelled as intervention group (recieving pre-operative music intervention), The group 2 will be labelled as controlled group (Not receiving pre-operative music intervention). Clinico-biochemical, Bio-cellular & Neurohumoral data evaluation will be done in both the groups.The results will be analyzed using standard SPSS software.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The Participants will be randomized to be part of the study groups. The Care providers will not be aware of the grouping of the participants as the intervention is done in the pre-operative holding area. All patients will undergo Laparoscopic Cholecystectomy under standard operative and anesthesia protocol. The Investigator (Nurse and the doctor staff) will also be unaware of the grouping of the patients. The recorded data will be analyzed by an individual outcome asser unaware of the grouping or identity of the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Experimental): Preoperative application of a Bluetooth enabled headphones with standard music played for atleast 2 hours preoperatively.
  Interventions: Other: Preoperative application of a bluetooth enabled Headphones.
- No Music (Active Comparator): Preoperative application of a Bluetooth enabled headphones with no music played and headphones will just mask the surrounding noise.
  Interventions: Other: Preoperative application of a bluetooth enabled Headphones.

INTERVENTIONS:
Other: Preoperative application of a bluetooth enabled Headphones. — A Bluetooth enabled Headphones device which is worn overhead and music can be played through it.

SUMMARY:
Surgery induced sterile inflammation leaves behind a biomolecular footprint measurable by various pro-inflammatory markers e.g. IL-6, CD(Cluster of differentiation)19B, HsCRP(High-sensitivity CRP) etc. Music is a non-pharmacological means in attenuating this inflammatory pathway thereby improving Health related quality of life measurable by improved postoperative convalescence. Correct timing of music application is a lacuna in the knowledge. This research aims at evaluating the effect of preoperative music on sterile inflammation induced by index Laparoscopic Surgery (Laparoscopic Cholecystectomy) and its proposed beneficial effects on patient reported outcomes. A total of 50 patients divided into 2 groups (test and control) will be evaluated in this triple blind randomized controlled study aiming at evaluating the biomolecular signatures of sterile inflammatory response and its correlation with improved postoperative convalescence. All the patients will be followed up for a period of 1 month postoperatively to assess for overall improvement in health related quality of life. Collected data will be analysed using updated SPSS software and a p value of less than 0.05 will be taken as statistically significant in support of the measured indices.

DETAILED DESCRIPTION:
INTRODUCTION Historically, surgery was seen as the last resort to preserve life. Even today, the popular acceptance of surgery is premised upon it being either as the only treatment option or as the last option after all nonsurgical treatments have been unsuccessful. This is attributable to the patient anxiety about the protracted convalescence, besides its clinical morbidity. Over last two centuries, surgery has evolved from being misery alleviating to being life-saving and then to being limb-preserving and finally function preserving as well. Last 30 years have witnessed the introduction of minimally invasive surgery (MIS) into surgical practice. Application of MIS in various surgical domains has achieved clinical equivalence with the established benchmarks of the conventional surgery. The spectrum of clinical equivalence besides positive outcomes includes the whole spectrum of the established various morbidity indicators like procedure specific complications, length of hospital stay and long-term morbidity. The focus for further evolution in surgery has marched from being clinical outcome based on the patient-reported outcome (PRO) specific. The improvement in PRO's has been attributed to attenuated postoperative inflammatory response, which has been studied by the changes in cytokine pathways. This cytokine-mediated inflammatory response is shown to be subdued after MIS as compared to conventional surgery.

Parallel to emphasis on PROs, surgery evolved with considerations for early and speedier convalescence. This led to the concept of enhanced recovery after surgery (ERAS) being the current stated objective. Postoperative convalescence (POC) is a function of the inflammatory response following surgery. This postoperative inflammatory response consists of a sterile inflammation apart from classical inflammation if any infection coexists. Sterile inflammation determines outcomes like postoperative fatigue (POF), postoperative pain (POP), postoperative nausea and vomiting (PONV) and circadian disturbances leading to compromised quality of sleep. All these factors directly influence postoperative convalescence as well as PROs. Patient perspective has been classically described by the aphorism "Surgery leaves scars on the mind as well". This sentiment now has scientific resonance, as now it is understood that the mediators of sterile inflammation are influenced temporarily and by neurohumoral pathways. Sterile inflammation is mediated by various cytokine and immunosuppressive pathways. It is primarily driven by danger associated molecular proteins (DAMP), also known as alarmins. These alarmins trigger a biocellular response by expansion of many cell lines. The CD19B cell line is known to expand the most. These biocellular responses then initiate a cascade of cytokines of which IL6 is the most dominant. It is the balance of these two, that determines the severity of sterile inflammation hence the POC. Current scientific discourse is on modulating this sterile inflammatory pathway. Pharmaceutical interventions by anti-inflammatory drugs are already known to attenuate this pathway and make the patient feel better but are not free of side effects. Non-pharmaceutical interventions have recently been studied for the same effect with an additional benefit of avoiding side effects of drugs. Perioperative music has been shown to improve both POC as well as PROs. However, this benefit has been reported for preoperative & peroperative music for surgeries under local or locoregional anaesthesia. Effect of preoperative music has not been studied for outcomes of surgeries done under general anaesthesia. The biocellular and biomolecular basis of this effect of music has not been clearly established. The most beneficial timing of music i.e. preoperative or peroperative is also not scientifically clear. The studies showing benefits of preoperative music are based upon surgeries under local-locoregional anaesthesia In a recent study done at our institution, study, peroperative music has been found to be beneficial. This study was done on the index MIS i.e. laparoscopic cholecystectomy (LC)under general anaesthesia (GA). Peroperative music was found to have a biocellular as well as biomolecular signature. It causes attenuation of sterile inflammation by controlling the expansion of CD19 cell population&, limiting the suppression of NK cell population and moderating the IL6 surge. Music-induced fall in IL6 as the beneficial biomolecular response has already been known.

With this background of established benefits of perioperative music but no study having tested preoperative music for surgery under GA, and an established known biocellular - biomolecular basis of peroperative / postoperative music for surgeries done under GA benefits, the investigator hypothesize that preoperative music could also have similar benefits for surgeries done under and GA, and a biomolecular basis for the same.

REVIEW OF LITERATURE Historically, practice of surgery started as the last resort for preservation of life. Over the last two centuries it has improved with progressive reduction in not only mortality but and significant improvements in clinical morbidity. With the advent of MIS, not only the clinical benchmarks of the conventional era were expected to be achieved matched with heightened community expectations. The practice of MIS was initially driven by its popular appeal despite the absence of any supportive level I evidence. The benefits of MIS were primarily based upon PROs. The benefits included reduced wound morbidity both in short-term (wound infections) as well as long-term (an incisional hernia). Other popular advantages included shorter hospital stay, less postoperative pain, lesser analgesia usage, early return to activity and better patient-reported health-related quality of life (HrQoL). All these made MIS popular both with society as well as with profession.

Application of MIS to most of the surgical domains was aided by paralleled advances in technological technology advances and innovations. In last 30 years of MIS experience, the clinical and PRO outcomes have stabilized. Current scientific discourse is on improving POC. Postoperative convalescence is akin to side effects of medicines in non-surgical practice. Postoperative convalescence is dependent upon various factors. Postoperative pain, PONV, POF, sleep disturbances and analgesia required are some of these factors. Postoperative convalescence is variable for similar surgeries. Prolonged POC leads to personal suffering, functional impairment, delayed return to work, and significant societal and economic costs. Postoperative convalescence has been defined as the "process to regain control over physical, psychological, social and habitual functions, and return to preoperative levels of independence and psychological well-being". It marks a shift from conventional recovery indicators e.g. length of hospital stay, to PROs like the absence of symptoms, the ability to perform regular activities, return to work, and regain quality of life. Major determinants of slow POC are fatigue, pain and resulting functional impairment. Fatigue is the key sickness behaviour fined as "an indefinable weakness throughout the body requiring sitting or lying down after minor tasks". The POC delaying factors are a clinical manifestation of an inflammatory process induced by surgery and stress of surgery. This inflammatory process happens in absence of any infective agent hence is called 'Sterile inflammation'. This sterile inflammation is a result of various cellular, biomolecular, immune changes induced by surgery. These are mediated by signalling that involves the production of cytokines, expansion of certain cell populations and contraction of some cell population. These changes happening within 24 hrs and are strongly associated with the speed of POC. Surgery induces a local immune response which leads to systemic proinflammatory and immunosuppressive phases which are temporally related and proportionate in magnitude. This response is mediated by a battery of cytokines of which IL6 is not only the beginner but also most dominant. Tissue injury is sensed by a group of protein receptors known as pattern recognition receptors (PRR). These PRRs can be activated by pathogen-associated molecular pattern (PAMP) and DAMP. The surgery induced sterile inflammation has no PAMP hence the DAMP is primary driver of the inflammatory cascade. Various pharmaceutical interventions (anti-inflammatory agents) have been used to attenuate or abort this sterile inflammation towards the goal of enhancing POC, but they are not free of side effects & contraindications. Music has been shown to have a positive influence on POC and PROs with supportive robust Level 1 evidence. Yet there is debate on many issues-

* Relative efficacy of preoperative music under general anaesthesia.
* Choice of music, whether patients or surgeons.
* Type of music, classical or otherwise.
* The timing of music, whether preoperative or peroperative or both.
* Whether patient alone or the entire OT team. These issues are pertinent because some surgeons accept the benefits to their patients but distracting to their staff. Some colleagues demand evidence better than the available Level 1 A evidence and consider it potential disruptor of communication& dangerous for patient safety. They find support from studies giving a scientific camouflage in concluding that music may contribute to decreasing in auditory processing function see music as noise in the OT. These naysayers have had robust rebuttals from other colleagues. Giving the choice of music to the patient has been shown to increase add to preoperative anxiety and compromise its benefits but some studies have advocated patient choice. But none of the studies has tested preoperative music for surgery done under GA. The investigator has earlier studied the effect of peroperative music and found it to be beneficial. It is not known whether preoperative music will have similar benefits or not? Hence, the investigator hypothesized to study this.

The benefits of music are related to attenuation of sterile inflammation and the inflammation is measurable with cytokine - immunosuppressive pathways. These pathways need to be studied for the effect of DAMPS. Thermal energy has a specific DAMP known case of heat called heat shock protein (HSP). The thermal energy specific sterile inflammation and its impact on PROs / POC have been reported earlier. This HSP related inflammatory component and its attendant cytokine response have also been studied and reported. As thermal component has its specific signature, any study of sterile inflammation induced by non-HSP DAMPs requires the surgery to be done without application of thermal energy. Hence an MIS procedure that is done without energy has to be subject to study. Laparoscopic cholecystectomy can be done safely, without an application of energized dissection by thermal energy. Laparoscopic cholecystectomy is an index MIS surgery for any innovations or PRO based studies.

A study of biomolecular changes and their effect on PROs, and POC in a setting of an HSP milieu, is thus an appropriate model to study the effect of preoperative music. Hence, the investigator proposes to study the biomolecular (IL6, TNF alpha, HSCRP, procalcitonin) and PROs (POP, PONV, POF, postoperative sleep quality, HrQoL and quantitative analgesia usage) in an HSP DAMP driven surgical milieu of an index MIS i.e. LC without the usage of surgical energy.

What is already known?

* Perioperative Peroperative and postoperative music are beneficial in improving 'postoperative convalescence' and 'patient reported outcomes' following surgery under all kinds of anaesthesia.
* These benefits are demonstrable in unaware (under GA) peroperative phase.
* The peroperative music related benefits have a quantitative biomolecular footprint.

Lacunae in our knowledge

* Effect of preoperative music on 'postoperative convalescence' and 'patient reported outcomes' following surgery under GA has not been studied.
* Biomolecular response specific to preoperative music in surgeries done even under locoregional anaesthesia (without GA) has not been studied.

HYPOTHESIS • Preoperative music could have beneficial effects on 'postoperative convalescence' and 'patient reported outcomes' following laparoscopic surgery under general anaesthesia GA.

AIMS AND OBJECTIVES

Primary objective:

• To study the effect of preoperative music on 'postoperative convalescence' and 'patient reported outcomes' following laparoscopic surgery under general anaesthesia'

Secondary objective:

• To study the biomolecular response specific to preoperative music.

MATERIALS AND METHODS

* STUDY SITE- Sir Ganga Ram Hospital, New Delhi.
* TIME & Duration of the study- From October 2017 until January 2019
* STUDY DESIGN-Triple-blinded Randomized Study
* SAMPLE SIZE - A reduction in pain scores (between 6-24 hours after surgery) from 48.04 (SD 11.07) to 26.54[16] (10.03) with a p-value of 0.000 has been seen in the investigator's previous study on the effect of peroperative music in the similar study population. To study the similar benefit of preoperative music with a confidence interval of 99% and an alpha error of 0.01 and power of 90%, a sample size of 16 i.e. 8 patients in each arm is required. With possible trial deviates attrition of 33%, the sample size required will be 24 (12 in each group). Given the window of time available, a minimum of 24 patients (12 in each group) but the desirability of population size similar to our last study with peroperative music, the investigator intends to have a sample size of 50 (25 in each group). An intention to treat analysis will be done.
* RANDOMIZATION- Computer generated randomization by an independent external research coordinator and will be telecommunicated to the nurse in preoperative area.

All participants found eligible and compliant with inclusion criteria will be enrolled for the study. Demographic and clinical data of the participants will be recorded in a standard proforma (Annexure II). A standard protocol for perioperative medicines including Anaesthesia, antibiotics, chemoprophylaxis and analgesia etc. will be followed.

The participants will be allocated to either study or control group by an independent external research co-coordinator (based upon a random sequence computer generation). The external coordinator will inform about the group allocation to the nurse in preoperative hold area (POHA), by phone or any web-based media network (SMS and/or WhatsApp).

A standard post-operative recovery clinical pathway compatible with ERAS and protocol for 'fast track surgery', will be followed by the discharge ability.

At the time of shifting of the patient, from the ward to POHA, a Bluetooth Headphone will be applied put on the participants. Once in POHA, an independent nurse will either start the music or not, as per the random group assigned. The participants will stay for 60 to 90 minutes in POHA. They will be shifted with the headphones to the operation theatre. The headphones will be removed at the time of induction of anaesthesia.

An EEG will be done in the ward before transfer to POHA, during surgery and 24 hours after surgery.

Blood samples will be drawn at the time of transfer from the ward to POHA i.e. prior to application of headphones (HT0), at the time of before induction of anaesthesia (TH1), at 6 hours after surgery (TH2) and at 24 hours after surgery (TH3).

• Premedication- All participants will receive premedication with alprazolam (0.25 mg) the night before surgery and ranitidine (150 mg per oral, the night before surgery and 120 min before surgery).

Anaesthesia Technique:

All participants will receive pre-induction fentanyl citrate 2 micrograms /kg. Routine monitoring (Pulse Oximetry, EKG, NIBP) will be applied. A bi-spectral index (BIS) sensor for monitoring the depth of Anaesthesia, using the BIS monitoring module, will also be applied over the participant's forehead according to the manufacturer's instructions prior to the induction of anaesthesia. After pre-oxygenation, anaesthesia will be induced with propofol up to 2.0mg/kg body weight to the point of loss of verbal contact. Atracurium besylate will be administered 0.5mg/kg to facilitate tracheal intubation. General Anaesthesia will be maintained with sevoflurane (1-2%) and 50% nitrous oxide in oxygen titrated to maintain a BIS value between 40-60. Fentanyl citrate 0.5 microgram/kg will be administered every 30 minutes intraoperatively.

Postoperatively, paracetamol 1 gm I.V. will be administered if the visual analogue scale (VAS) score is >30.

The hemodynamic markers of the depth of Anaesthesia like pulse, blood pressure, saturation of peripheral oxygen (SpO2), and end-tidal carbon dioxide (EtCO2) concentration will be recorded in a standard proforma (Annexure III). Standard four-port technique of LC without energized dissection will be followed [35].

The surgical procedure will be video-recorded for prospective anatomical analysis and retrospective reference. Duration of surgery will be recorded with reference to the different stations of intervention i.e. induction of anaesthesia, first surgical incision, complete separation of GB from liver bed and extubation. Peroperative surgical data will be recorded in a standard proforma.

Operative clinical data will be recorded in a standard proforma. This post-operative protocol will be followed by the surgical nurses in the common post-operative area where all the operated cases are managed. Standard criteria based discharged protocol will be followed.

Participants will be discharged after clearance from with protocol-based consensus of the anaesthesia team, nursing team and surgical team. A standard discharge advice will be given to the participants incorporating the various post-operative diary protocols.

The PRO's and the clinical outcome will be analyzed by Clavien and Dindo classification of surgical complication.

Statistical Analysis The prospectively collected data will be entered into an excel sheet (Windows Microsoft 8 or higher version). The data will be analyzed using the latest version of SPSS (statistical package for social science). Qualitative data will be compared using Chi-square test and quantitative data using Student's t-test, or any other appropriate statistical tool. A p-value less than 0.05 will be considered significant. An intention to treat analysis will be done.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 18 years.
2. Should be able to understand and sign an informed consent.
3. Consent for surgery, anaesthesia and the use of standardized music before surgery. (Appendix I)
4. Fitness for General Anesthesia (GA)
5. Ability to maintain & communicate a PRO diary.
6. Ability to communicate via telephone or email or SMS or WhatsApp.

Exclusion Criteria:

1. Fitfor GA but higher than ASA Grade I.
2. Uncontrolled coagulopathy
3. Suspicion of carcinoma gallbladder on USG
4. Any suspicion of common bile duct (CBD) stones or pancreatitis.
5. Patient using chronic anti-inflammatory drug.
6. Concomitant common bile duct (CBD) stone or any CBD intervention/pancreatitis in the preceding 6 weeks.
7. Patient on immunosuppressive / cytotoxic/ steroid therapy.
8. Documented or known sensitivity to any drug to be used in the study protocol.
9. Pregnant or lactating ladies.
10. Any concomitant surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain (POP) | 3 weeks
  Visual Analogue Scale (VAS) will be used to measure the pain on a numeric scale of 0-100 at 6 Hours, Day 1, Day 3, Day 10 and Week 3 postoperatively respectively with a total of 5 readings. Higher values on the VAS will represent a worse outcome.
  Minimum value on VAS = 0 Maximum value on VAS= 100
Postoperative Nausea Vomiting (PONV) | 3 weeks
  Visual Analogue Scale (VAS) will be used to measure the PONV on a numeric scale of 0-100 at 6 Hours, Day 1, Day 3, Day 10 and Week 3 postoperatively respectively with a total of 5 readings. Higher values on the VAS will represent a worse outcome.
  Minimum value on VAS = 0 Maximum value on VAS= 100
Postoperative Fatigue (POF) | 3 weeks
  Visual Analogue Scale (VAS) will be used to measure the pain on a numeric scale of 0-100 at 6 Hours, Day 1, Day 3, Day 10 and Week 3 postoperatively respectively with a total of 5 readings. Higher values on the VAS will represent a worse outcome.
  Minimum value on VAS = 0 Maximum value on VAS= 100
Gastrointestinal Quality of Life Index (GIQoL) | 1 month
  Gastrointestinal Quality Of Life Index (GIQoL) 30 Days Min=0 (Best) Max=144 (Worst) GIQoL will be assessed on 30th postoperative day and any difference in the measurement will be assessed for analysis in between the two study arms.

SECONDARY OUTCOMES:
Liver function test (LFT) | upto 24 hours after surgical intervention
  Tests will be done for 4 times (Preoperatively, Intraoperatively, 6 hours postoperatively, 24 hours postoperatively)
Serum amylase | upto 24 hours after surgical intervention
  Tests will be done for 4 times (Preoperatively, Intraoperatively, 6 hours postoperatively, 24 hours postoperatively)
  The difference in the values will be assessed as follows for all the testes:
  Preop-Intraop, Intraop-6H, 6H-24H
Serum lipase | upto 24 hours after surgical intervention
  Tests will be done for 4 times (Preoperatively, Intraoperatively, 6 hours postoperatively, 24 hours postoperatively)
  The difference in the values will be assessed as follows for all the testes:
  Preop-Intraop, Intraop-6H, 6H-24H
Interlukin-6 (IL-6) | upto 24 hours after surgical intervention
  Tests will be done for 4 times (Preoperatively, Intraoperatively, 6 hours postoperatively, 24 hours postoperatively)
  The difference in the values will be assessed as follows for all the testes:
  Preop-Intraop, Intraop-6H, 6H-24H
Tumor Necrosis Factor-alpha (TNF -alpha ) | upto 24 hours after surgical intervention
  Tests will be done for 4 times (Preoperatively, Intraoperatively, 6 hours postoperatively, 24 hours postoperatively)
  The difference in the values will be assessed as follows for all the testes:
  Preop-Intraop, Intraop-6H, 6H-24H
HsCRP | upto 24 hours after surgical intervention
  Tests will be done for 4 times (Preoperatively, Intraoperatively, 6 hours postoperatively, 24 hours postoperatively)
  The difference in the values will be assessed as follows for all the testes:
  Preop-Intraop, Intraop-6H, 6H-24H
Serum Procalcitonin | upto 24 hours after surgical intervention
  Tests will be done for 4 times (Preoperatively, Intraoperatively, 6 hours postoperatively, 24 hours postoperatively)
  The difference in the values will be assessed as follows for all the testes:
  Preop-Intraop, Intraop-6H, 6H-24H
EEG | upto 24 hours after surgical intervention
  Recording of EEg will be done at 3 separate occasions. Preoperatively, Intraoperatively and 24 hours postoperatively. EEG will be interpreted by a an independent evaluator for any changes who will be unaware of the timing of record of the EEG. The changes in the brain wave form will be seen and recorded for evaluation.
LDH | upto 24 hours after surgical intervention
  Tests will be done for 4 times (Preoperatively, Intraoperatively, 6 hours postoperatively, 24 hours postoperatively)
  The difference in the values will be assessed as follows for all the testes:
  Preop-Intraop, Intraop-6H, 6H-24H
Uric Acid | upto 24 hours after surgical intervention
  Tests will be done for 4 times (Preoperatively, Intraoperatively, 6 hours postoperatively, 24 hours postoperatively)
  The difference in the values will be assessed as follows for all the testes:
  Preop-Intraop, Intraop-6H, 6H-24H

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Brij Bushan Agarwal, Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided
Clinical and biochmical data